CLINICAL TRIAL: NCT02257229
Title: Prospective Evaluation of Treatment for Clubfoot
Status: Recruiting | Type: Observational
Sponsor: Texas Scottish Rite Hospital for Children (Other)
Responsible Party: Principal Investigator, Anthony Riccio, Principal Investigator, Texas Scottish Rite Hospital for Children
Other Study IDs: 032011-131
Record Dates: First submitted 2014-09-22; First posted 2014-10-06 (Estimated); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Clubfoot Deformity
Keywords: Clubfoot, deformity, correction, management, gait
MeSH Terms: conditions — Clubfoot; Congenital Abnormalities | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Surgical: Corrective Surgery only
  Interventions: Procedure: Surgical
- Non-Surgical: Correction with casting, braces, Physical therapy, other non-surgical methods
  Interventions: Procedure: Non-Surgical
- Non-surgical + surgical: Correction with casting, braces, Physical therapy, other non-surgical methods subsequently followed by Corrective Surgery
  Interventions: Procedure: Non-surgical + surgical

INTERVENTIONS:
Procedure: Surgical — Surgery only
  Groups: Surgical
Procedure: Non-Surgical — non-surgical methods such as, casting, bracing, physical therapy, and other.
  Groups: Non-Surgical
Procedure: Non-surgical + surgical — Combination of non-surgical methods subsequently followed by surgery
  Groups: Non-surgical + surgical

SUMMARY:
Specific aim:

To evaluate the outcome of infants who undergo one of two nonsurgical treatment interventions

DETAILED DESCRIPTION:
PURPOSE: The purpose of this project is to help orthopaedic surgeons better understand and treat patients with a diagnosis of clubfoot. This proposed research will establish a protocol for the collection of relevant clinical and functional outcome measures on our patients with a diagnosis of clubfoot.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of clubfoot deformity
* Spanish speaking patients will be eligible to participate in the study.

Exclusion Criteria:

* All patients without a diagnosis of clubfoot

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2005-08; Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Degree of correction at initial brace wear | 2 months
  Dimeglio scoring system will be used (score range from 0-20)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony I Riccio, MD, Principal Investigator — Texas Scottish Rite Hospital for Children
Locations (1):
- Texas Scottish Rite Hospital for Children, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Data will be collected at one site, only results of data analysis will be release in publishing. Data itself will not be shared.